CLINICAL TRIAL: NCT00272064
Title: Optimisation of Insulin Treatment of Type 2 Diabetes Mellitus by Telecare Assistance for Self Monitoring of Blood Glucose (SMBG).
Brief Title: ELEONOR STUDY: Insulin Glulisine in Type 2 Diabetes Mellitus.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMR1964A_3514; EudraCT # : 2004-002731-62
Record Dates: First submitted 2006-01-02; First posted 2006-01-04 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin glulisine; Insulin Glargine; Metformin

ARMS (2):
- 1 (Other): Telecare system
  Interventions: Drug: Insulin glulisine; Drug: Insulin glargine; Drug: Metformin
- 2 (Other): Self Monitoring Blood Glucose (SMBG)system.
  Interventions: Drug: Insulin glulisine; Drug: Insulin glargine; Drug: Metformin

INTERVENTIONS:
Drug: Insulin glulisine — individualized, once daily, dose aiming at 2h post-prandial plasma glucose goal < 140 mg/dl (7.8 mmol/l) in the optimized treatment phase, since visit 3, subcutaneous
Drug: Insulin glargine — individualized, once daily, dose to reach mean fasting plasma glucose (FPG) <= 126 mg/dl (7.0 mmol/l), since randomization, subcutaneous
Drug: Metformin — 1000 mg b.i.d, since the qualification phase, oral

SUMMARY:
* The primary objective of the present study is to verify the superiority of Telecare program vs. standard SMBG program in terms of mean HbA1c value (- 0,5%) at end-point.
* The secondary objectives of the study are the assessment of: total daily dose of insulin, changes in glycaemic and lipid profile, frequency of hypoglycaemias, changes in weight, health-related quality of life, cost-effectiveness of Telecare program vs. common ambulatory program; general safety (adverse event profile, other routine laboratory parameters).

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of type 2 Diabetes Mellitus
* Patients treated with combined oral antidiabetic drugs(as fixed combination or simultaneous administration) or with metformin in monotherapy at maximal doses for at least 3 months
* Patients having BMI > 25 Kg/m2;
* Patients having a HbA1c ≥ 7.5 % and ≤ 11 %
* Female patients must be menopausal, surgically sterile, or using effective contraceptive measures;
* Female of childbearing potential must use effective contraceptive measures for at least 1 month prior to the entry into the study and should continue to use the same contraceptive method during the overall study period.

Exclusion criteria:

* Patients diagnosed with type 1 insulin dependent Diabetes Mellitus;
* History of two or more severe hypoglycaemic episodes within the past 3 months or history of unawareness hypoglycaemia;
* Active proliferative diabetic retinopathy, as defined by the application of focal or panretinal photocoagulation or vitrectomy, in the 6 months prior to visit 1, or any other unstable (rapidly progressing) retinopathy that may require surgical treatment (including laser photocoagulation);
* Impaired renal function
* Impaired liver function
* History of hypersensitivity to insulin or insulin analogues or any of the excipients in the Insulin glulisine and Insulin glargine formulation
* History of hypersensitivity to metformin;
* Pregnant or breast-feeding women, or women planning to become pregnant during the study;
* Failure to use adequate contraception (women of current reproductive potential only);
* Any clinically significant major organ system disease such as relevant cardiovascular, gastrointestinal, hepatic, neurological, endocrine, haematological or other major systemic diseases or infective diseases;
* History of drug or alcohol abuse within the last 2 years or current addiction to substances of abuse;
* Night shift workers;
* Receipt of an experimental drug or use of an experimental device within the 30 days prior to study entry;
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study;
* Treatment or likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol;
* Any disease or condition including abuse of illicit drugs, prescription medicines or alcohol that in the opinion of the investigator or sponsor may interfere with the completion of the study;
* Subject unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study procedures;
* Subject is the investigator or any sub investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol;
* Previous enrolment in the present study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2005-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Changes of glycosilated haemoglobin (HbA1c) | At least 12 weeks from baseline (visit 3)

SECONDARY OUTCOMES:
Changes in fasting plasma glucose | At each visit
Changes in plasma insulin levels | At each visit
Change of Self-monitoring of Blood Glucose (SMBG) | for the total study duration
Mean Amplitude Glucose Excursion (MAGE) | for the total study duration
Change in lipid profile | V1 (screening) and V5 (end of treatment)
Body weight - Body Mass Index | V1 (screening), V3 (start of titration), V4 (after 12 weeks of treatment), V5 (end of treatment), V6 (end of follow-up)
Total daily dose of insulins (glargine and glulisine) | At each visit (starting from V2 for glargine and from V3 for glulisine)
Health related Quality of Life | V2 (start of titration), V4 (after 12 weeks of treatment), V5 (end of treatment)
Hypoglycemic episodes | for the total study duration

CONTACTS AND LOCATIONS:
Overall Officials: PAIZIS GEORGES, MD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Milan, Italy

REFERENCES:
- [Derived] Del Prato S, Nicolucci A, Lovagnini-Scher AC, Turco S, Leotta S, Vespasiani G; ELEONOR Study Group. Telecare Provides comparable efficacy to conventional self-monitored blood glucose in patients with type 2 diabetes titrating one injection of insulin glulisine-the ELEONOR study. Diabetes Technol Ther. 2012 Feb;14(2):175-82. doi: 10.1089/dia.2011.0163. Epub 2011 Oct 20. PMID 22013886